CLINICAL TRIAL: NCT02492906
Title: Neuroimaging of Patients With Severe Knee Osteoarthrosis - Evaluation of Cerebral Volumetry
Status: Completed | Type: Observational
Sponsor: Marta Imamura (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, Coordinator of the Clinical Research Site of Institute of Physical and Rehabilitation Medicine of HC FMUSP, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: Osteoarthrosis Neuroimaging
Record Dates: First submitted 2015-06-29; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — ORALIT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Osteoarthrosis group: Patients with primary severe knee osteoarthrosis or with chronic knee pain.
  Interventions: Other: Osteoarthrosis
- Healthy patients: Healthy patients
  Interventions: Other: Healthy

INTERVENTIONS:
Other: Osteoarthrosis — Primary severe knee osteoarthrosis and chronic knee pain.
  Groups: Osteoarthrosis group
Other: Healthy — Healthy and non-symptomatic volunteers.
  Groups: Healthy patients

SUMMARY:
Due to scarce published articles about this subject, the researchers aim to study the volume measurements of the brain cortex of patients with primary severe knee osteoarthrosis and those with chronic knee pain compared to healthy and non-symptomatic volunteers, correlating the neuroimaging of cerebral volumetry with pain intensity, pain duration, knee function and pressure pain threshold.

DETAILED DESCRIPTION:
The protocol was designed to include 31 patients in each observational arm, either patients with severe knee osteoarthrosis and chronic knee pain or healthy and non-symptomatic volunteers.

The researchers performed anamnesis to collect clinical and demographic information, the intensity of pain was assessed by the self-rated Visual Analogue Scale (VAS), the pressure pain threshold was evaluated with an algometer, the knee function was assessed with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale and the images were collected with the use of the Magnetic Resonance.

Covariates, such as age, gender, Body Mass Index (BMI) and comorbidities as diabetes, cardiac diseases, pulmonary diseases, endocrine diseases and the practice of physical activities were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years old;
* Both genders;
* Clinical diagnosis of knee osteoarthrosis;
* Self-rated VAS moderate to severe (VAS > 4);
* Pain duration longer than 3 months prior to the evaluation;
* Signed Informed Consent;
* Light physical activity practice or sedentary (healthy volunteers only).

Exclusion Criteria:

* Presence of psychiatric disorders;
* Presence of fibromyalgia;
* Presence of rheumatologic diseases;
* Presence of previous knee surgery;
* Presence of clinical symptoms (healthy volunteers only);
* Presence of knee pain on the previous 6 months (healthy volunteers only);
* History of neoplasia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients and patients with primary severe knee osteoarthrosis and with chronic knee pain were included.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cerebral Volumetry Comparison | Baseline at time of evaluation.
  Brain Magnetic Resonance on axial Fluid Attenuated Inversion Recovery (FLAIR) and axial volume comparison between the healthy and the Knee Osteoarthrosis Group.

SECONDARY OUTCOMES:
VAS Comparison | Baseline at time of evaluation.
  Self rated Visual Analogue Scale for pain comparison between the healthy and the Knee Osteoarthrosis Group.
Pressure Pain Threshold Comparison | Baseline at time of evaluation.
  Pressure algometry on the patients' back and lower limbs for comparison between the healthy and the Knee Osteoarthrosis Group.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, São Paulo, Brazil